CLINICAL TRIAL: NCT00417508
Title: Effectiveness of Nutritional Intervention in Malnourished Elderly Patients
Brief Title: Nutritional Intervention in Malnourished Elderly Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: It was not possible to recruite sufficient number of participants
Sponsor: University Hospital of North Norway (Other)
Collaborators: Centre for Research in the Elderly, Tromsoe, Norway (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P REK NORD 64/2003
Record Dates: First submitted 2006-12-29; First posted 2007-01-01 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2012-06

CONDITIONS: Malnutrition
Keywords: function; elderly; ADL; nutritional supplementation; Quality of life; handgrip strength; Body Composition
MeSH Terms: conditions — Malnutrition | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional supplement (Experimental): 2 packages/day with nutritional supplement containing a total of 600 kcal and 40 g protein
  Interventions: Dietary Supplement: Sip feeding
- Dietary advice (Active Comparator): ordinary dietary advice with a recommendation of four meals per day or similar dietary advice
  Interventions: Dietary Supplement: Dietary Advice

INTERVENTIONS:
Dietary Supplement: Sip feeding — Daily supplement with sip feeding, 2 packages(each package containing 200 ml,20 g protein and 300 kcal)
  Other Names: Fresubin Protein Energy Drink
  Arms: Nutritional supplement
Dietary Supplement: Dietary Advice — The patients will receive ordinary dietary advice with a recommendation of four meals per day or similar dietary advice and no daily sip feeding supplements.
  Arms: Dietary advice

SUMMARY:
The purpose of this study is to investigate whether nutritional supplementation will improve functional outcome parameters and nutritional status in elderly patients.

DETAILED DESCRIPTION:
Malnutrition is still a problem in elderly patients and this may be associated with reduced muscle strength and ADL function (activities of daily living). Malnourished Medical Inpatients/Outpatients and District Nurse patients with a Body Mass Index < 20 kg/m2 are asked to participate.

Comparison(s): The patients are randomized to either ordinary dietary advice with a recommendation of four meals per day or similar dietary advice and two daily sip feeding supplements. The study supplementation is Fresubin Protein Energy Drink and this will give additional 600 kcal and 40 gram protein a day. The study period is 12 weeks with a visit at inclusion, week 6 and week 12.

Primary and secondary outcome parameters are measured at inclusion and week 12

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index < 20 kg/m2
* Medical In/Outpatient or District Nurse-patient
* Able to take nutritional supplement (sip feeding)
* Able to walk
* Written patient informed consent

Exclusion Criteria:

* Actual malignancy
* Dementia with a Mini Mental Status score < 24
* Severe depression
* Need for Total Parenteral Nutrition or Tube Feeding
* Prescribed nutritional supplements during more than the last week
* Life expectancy of less than 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Functional Health (Short form 36) | Start and 12 weeks

SECONDARY OUTCOMES:
Nutritional Measures (at inclusion and week 12) | Start and 12 weeks
Change in Body weight and Lean Body Mass(evaluated with dual energy X-ray absorptiometry) | at 6 and 12 weeks
Psychological Measures (at inclusion and week 12) Hospital Anxiety and Depression scale | Start and 12 weeks
Observed ADL | Start and at 12 weeks
  Barthels index
Timed Up and Go test | Start and12 weeks
Hand grip strength | Start and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jon R Florholmen, MD, PhD, Study Chair — University Hospital of Northern Norway, Dep of Medical Gastroenterology
Locations (1):
- University Hospital of Northern Norway, Dep of Medical Gastroenterology, Tromsø, Tromsoe, Norway